CLINICAL TRIAL: NCT00975078
Title: Dexamethasone-suppression-test Predicts Later Development of Adrenal Insufficiency After a 14 Days' Course of Prednisone in Healthy Volunteers
Brief Title: Test Predicting Adrenal Insufficiency in Volunteers Under Prednisone Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Mirjam Christ-Crain, Endocrinology, University Hospital Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DEXA
Record Dates: First submitted 2009-09-07; First posted 2009-09-11 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Adrenal Gland Hypofunction
Keywords: dexamethasone-suppression-test; high dose glucocorticoid treatment; Population at Risk
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adrenal insufficiency (Experimental)
  Interventions: Procedure: adrenal insufficiency testing; Drug: prednisone

INTERVENTIONS:
Procedure: adrenal insufficiency testing — On the day getting the baseline data we will perform a low dose cosyntropin test to asses adrenal axis function.
  All participants will then undergo an overnight 0.5mg dexamethasone suppression test. Thereby participants will take 0.5mg of dexamethasone at 11 pm and a fasting blood sample will be collected the next morning at 8 am to measure the serum cortisol level.
  Six days later participants will start taking 0.5mg/kg body-weight prednisone each morning for 14 days.
  On day 1, 3, 7 and 21 after withdrawal of prednisone the participant will undergo a low dose cosyntropin test. The investigators will take a blood sample before and 30 minutes after i.v. administration of 1ug of cosyntropin for the measurement of cortisol.
Drug: prednisone — 0.5mg/kg body-weight prednisone each morning for 14 days

SUMMARY:
Suppression of the adrenal function is a common, potentially dangerous and unpredictable consequence of short term high dose glucocorticoid treatment. Identification of patients at risk would be of high clinical importance. The investigators hypothesized that the dexamethasone-suppression-test predicts the subsequent development of corticosteroid induced adrenal insufficiency.

DETAILED DESCRIPTION:
The objective of this study is to evaluate if adrenal axis integrity investigated by the dexamethasone-suppression-test will predict the development of adrenal insufficiency after 14 days treatment with 0.5mg/kg of body weight prednisone in healthy volunteers. The investigators hypothesize that subjects with a more suppressed cortisol level after dexamethasone will be more likely to develop adrenal insufficiency after 14 days intake of prednisone o.5mg/kg/body weight than subjects with less suppression of their cortisol levels after dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers over 18 years

Exclusion Criteria:

* No informed consent
* Intake of any kind of medication
* BMI over 30kg/m2
* Acute or chronic illnesses

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is the rate of adrenal insufficiency assessed on the 7th day after stopping a 14-days course of corticosteroid therapy with 0.5mg/kg KG prednisone per day. | 7th day after stopping prednisone intake

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Professor, Principal Investigator — Division of Endocrinology University Hospital Basel
Locations (1):
- Division of Endocrinology University Hospital Basel, Basel, Basel, Switzerland